CLINICAL TRIAL: NCT02460978
Title: A Multicenter, Randomized, Double-Blind, Placebo-controlled, Parallel Group, Phase 3 Study to Evaluate the Efficacy and Safety of Dapagliflozin as an Add-on to Insulin Therapy in Subjects With Type 1 Diabetes Mellitus - Study Two
Brief Title: Dapagliflozin Evaluation in Patients With Inadequately Controlled Type 1 Diabetes
Acronym: DEPICT 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB102-230; 2014-004599-49 (EudraCT Number); D1695C00007 (Other: AstraZeneca)
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Results first posted 2018-11-06 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Dapagliflozin; Efficacy; Safety; Add on to insulin; Oral Antidiabetic; Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dapagliflozin 5 mg (Experimental): Dapagliflozin 5 mg tablet orally, once daily for 52 weeks
  Interventions: Drug: Dapagliflozin
- Dapagliflozin 10 mg (Experimental): Dapagliflozin 10 mg tablet orally, once daily for 52 weeks
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo tablet orally, once daily for 52 weeks
  Interventions: Other: Placebo for dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Tablets
  Arms: Dapagliflozin 10 mg; Dapagliflozin 5 mg
Other: Placebo for dapagliflozin — Tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if adding dapagliflozin to insulin is a safe and effective therapy to improve glycemic control in patients with type 1 diabetes.

DETAILED DESCRIPTION:
Study Classification: Safety, Efficacy and Pharmacokinetics/dynamics

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 Diabetes mellitus (T1DM)
* Central laboratory C-peptide < 0.7 ng/ml (0.23 nmol/L)
* Insulin use for at least 12 months per patient reported or medical records
* Method of insulin administration (MDI or CSII) must have been unchanged for at least 3 months prior to screening
* Subjects must be on a total insulin dose of ≥ 0.3 U/kg/day for at least 3 months prior to screening
* If on MDI insulin administration, subject must be on ≥ 3x injections per day
* Screening Visit: Central laboratory HbA1c ≥ 7.7% and ≤ 11.0%
* Body mass index (BMI) ≥ 18.5 kg/m2

Exclusion Criteria:

* History of Type 2 Diabetes mellitus (T2DM) or maturity onset diabetes of the young (MODY), pancreatic surgery, or chronic pancreatitis that could result in decreased beta cell capacity
* Taking any non-insulin antihyperglicemic agent within 1 month prior to screening
* Taking GLP-1 receptor agonist within 2 months prior to screening for once weekly administration and within 1 month prior to screening for once or twice daily administration
* Taking metformin and/or thiazolidinediones within 2 months prior to screening
* History of diabetes ketoacidosis requiring medical intervention within 1 month prior to screening
* History of hospital admission for glycemic control (either hyperglycemia or hypoglycemia) within 1 month prior to screening
* Frequent episodes of severe hypoglycemia (more than one episode requiring medical assistance, emergency care), and/or glucagon therapy administered by a third-party individual within 1 month prior to screening
* History of Addison's disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 815 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2017-09-02 (Actual); Study Completion 2018-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Langkilde, MD, Study Director — AstraZeneca
Locations (123):
- United States (43):
  - Research Site, Concord, California
  - Research Site, Fresno, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, San Mateo, California
  - Research Site, San Ramon, California
  - Research Site, Walnut Creek, California
  - Research Site, Golden, Colorado
  - Research Site, Newark, Delaware
  - Research Site, Bradenton, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Springs, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Roswell, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Des Moines, Iowa
  - Research Site, Overland Park, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Kalamazoo, Michigan
  - Research Site, Edina, Minnesota
  - Research Site, Jefferson City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Reno, Nevada
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, Flushing, New York
  - Research Site, Mineola, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Amarillo, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Edinburg, Texas
  - Research Site, Mesquite, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Bennington, Vermont
  - Research Site, Federal Way, Washington
- Argentina (6):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Mar del Plata
  - Research Site, Ramos Mejía
- Belgium (2):
  - Research Site, Brussels (Uccle)
  - Research Site, Leuven
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Halifax, Nova Scotia
  - Research Site, Cambridge, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Smiths Falls, Ontario
  - Research Site, Sherbrooke, Quebec
- Chile (2):
  - Research Site, Santiago
  - Research Site, Temuco
- Germany (11):
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Falkensee
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Oldenburg
  - Research Site, Pohlheim
  - Research Site, Saarlouis
  - Research Site, Sulzbach-Rosenberg
  - Research Site, Wangen
- Japan (28):
  - Research Site, Aki-gun
  - Research Site, Amagasaki-shi
  - Research Site, Chitose-shi
  - Research Site, Chūōku
  - Research Site, Fukuyama-shi
  - Research Site, Higashiosaka-shi
  - Research Site, Ibusuki-shi
  - Research Site, Kagoshima
  - Research Site, Kamakura-shi
  - Research Site, Kashiwara-shi
  - Research Site, Kitakyushu-shi
  - Research Site, Koriyama-shi
  - Research Site, Kumamoto
  - Research Site, Kurume-shi
  - Research Site, Miura-shi
  - Research Site, Nagoya
  - Research Site, Obihiro-shi
  - Research Site, Osaka
  - Research Site, Oyama-shi
  - Research Site, Ōita
  - Research Site, Sapporo
  - Research Site, Shibuya-ku
  - Research Site, Shinjuku-ku
  - Research Site, Shizuoka
  - Research Site, Tsukuba
  - Research Site, Ushiku-shi
  - Research Site, Uwajima-shi
  - Research Site, Yokohama
- Netherlands (3):
  - Research Site, Hoogeveen
  - Research Site, Maastricht
  - Research Site, Utrecht
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (2):
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
- Sweden (4):
  - Research Site, Gothenburg
  - Research Site, Helsingborg
  - Research Site, Linköping
  - Research Site, Uddevalla
- Switzerland (3):
  - Research Site, Olten
  - Research Site, Sankt Gallen
  - Research Site, Zollikerberg
- United Kingdom (5):
  - Research Site, Manchester
  - Research Site, Northampton
  - Research Site, Oldham
  - Research Site, Swansea
  - Research Site, Wakefield

REFERENCES:
- [Derived] Nardone M, Kugathasan L, Sridhar VS, Dutta P, Campbell DJT, Layton AT, Perkins BA, Barbour S, Lam TKT, Levin A, Lovblom LE, Mucsi I, Rabasa-Lhoret R, Rac VE, Senior P, Sigal RJ, Stanimirovic A, Persson F, Stougaard EB, Doria A, Cherney DZI. Modeling Cardiorenal Protection with Sodium-Glucose Cotransporter 2 Inhibition in Type 1 Diabetes: An Analysis of DEPICT-1 and DEPICT-2. Clin J Am Soc Nephrol. 2025 Apr 1;20(4):529-538. doi: 10.2215/CJN.0000000641. Epub 2025 Feb 7. PMID 39918875
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Melin J, Tang W, Rekic D, Hamren B, Penland RC, Boulton DW, Parkinson J. Dapagliflozin Pharmacokinetics Is Similar in Adults With Type 1 and Type 2 Diabetes Mellitus. J Clin Pharmacol. 2022 Oct;62(10):1227-1235. doi: 10.1002/jcph.2062. Epub 2022 May 2. PMID 35403243
- [Derived] Groop PH, Dandona P, Phillip M, Gillard P, Edelman S, Jendle J, Xu J, Scheerer MF, Thoren F, Iqbal N, Repetto E, Mathieu C. Effect of dapagliflozin as an adjunct to insulin over 52 weeks in individuals with type 1 diabetes: post-hoc renal analysis of the DEPICT randomised controlled trials. Lancet Diabetes Endocrinol. 2020 Oct;8(10):845-854. doi: 10.1016/S2213-8587(20)30280-1. PMID 32946821
- [Derived] Mathieu C, Dandona P, Birkenfeld AL, Hansen TK, Iqbal N, Xu J, Repetto E, Scheerer MF, Thoren F, Phillip M. Benefit/risk profile of dapagliflozin 5 mg in the DEPICT-1 and -2 trials in individuals with type 1 diabetes and body mass index >/=27 kg/m2. Diabetes Obes Metab. 2020 Nov;22(11):2151-2160. doi: 10.1111/dom.14144. Epub 2020 Aug 20. PMID 32691513
- [Derived] Parkinson J, Tang W, Astrand M, Melin J, Ekholm E, Hamren B, Boulton DW. Model-based characterization of the relationship between dapagliflozin systemic exposure and HbA1c response in patients with type 1 diabetes mellitus. Diabetes Obes Metab. 2019 Jun;21(6):1381-1387. doi: 10.1111/dom.13664. Epub 2019 Mar 14. PMID 30756462
- [Derived] Mathieu C, Dandona P, Gillard P, Senior P, Hasslacher C, Araki E, Lind M, Bain SC, Jabbour S, Arya N, Hansen L, Thoren F, Langkilde AM; DEPICT-2 Investigators. Efficacy and Safety of Dapagliflozin in Patients With Inadequately Controlled Type 1 Diabetes (the DEPICT-2 Study): 24-Week Results From a Randomized Controlled Trial. Diabetes Care. 2018 Sep;41(9):1938-1946. doi: 10.2337/dc18-0623. Epub 2018 Jul 19. PMID 30026335
- See also: MB102230_CSP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4122&filename=MB102230_CSP.pdf
- See also: MB102230_SAP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4122&filename=MB102230_SAP.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The results on this form are from the 24 week short-term double-blind treatment period. This study was conducted at 148 centers in 13 countries from 8 July 2015 to 2 Sep 2017.
Pre-assignment Details: 815 participants were randomized. Of the 195 participants not randomized: 97 No longer met study criteria, 44 withdrew consent, 13 were lost to follow-up, and 41 did not continue for other reasons. Two participants did not receive any study drug and were excluded from analyses. Thus, the total number of subjects is 813.
Groups:
- DAPA 5 MG + INS: Dapagliflozin 5 mg plus insulin
- DAPA 10 MG + INS: Dapagliflozin 10 mg plus insulin
- PLA + INS: Placebo plus insulin
Period: Overall Study
Arm/Group | DAPA 5 MG + INS | DAPA 10 MG + INS | PLA + INS
Started | 271 | 270 | 272
Completed | 244 | 245 | 239
Not Completed | 27 | 25 | 33
Not completed — Adverse Event | 17 | 11 | 11
Not completed — Withdrawal by Subject | 5 | 5 | 14
Not completed — Lost to Follow-up | 2 | 3 | 1
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Discontinued due to DKA/hypoglycemia | 2 | 5 | 4
Not completed — Pregnancy | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DAPA 5 MG + INS | DAPA 10 MG + INS | PLA + INS | Total
Number analyzed (Participants) | 271 | 270 | 272 | 813
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.7 (13.35) | 42.4 (12.80) | 43.0 (13.73) | 42.7 (13.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 149 | 153 | 455
  Male | 118 | 121 | 119 | 358
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 210 | 219 | 208 | 637
  Black or African-American | 4 | 7 | 1 | 12
  Asian | 57 | 44 | 59 | 160
  Other | 0 | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in HbA1c at Week 24
Description: To compare the change from baseline in HbA1c between dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
Time Frame: Baseline and 24 weeks
Population: The analysis population for this endpoint is the number of subjects in the full analysis set with non-missing baseline and at least one post-baseline value. The full analysis set consists of all randomized subjects who took at least one dose of double-blind study medication during the short-term double-blind period.
Measure: Least Squares Mean (95% Confidence Interval); unit: HbA1c (%)
Arm/Group | DAPA 5 MG + INS | DAPA 10 MG + INS | PLA + INS
Number analyzed (Participants) | 266 | 267 | 267
HbA1c (%) | -0.34 [-0.43 to -0.25] | -0.39 [-0.48 to -0.30] | 0.03 [-0.06 to 0.12]
Statistical Analysis 1: Comparison: DAPA 5 MG + INS vs PLA + INS; Difference vs. placebo in adjusted mean change from baseline; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Model is adjusted for baseline HbA1c, treatment, week, randomization stratum, week*treatment, and week*baseline HbA1c; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.49 to -0.26], Standard Error of Mean 0.0579
Statistical Analysis 2: Comparison: DAPA 10 MG + INS vs PLA + INS; Difference vs. placebo in adjusted mean change from baseline; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Model is adjusted for baseline HbA1c, treatment, week, randomization stratum, week*treatment, and week*baseline HbA1c; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.53 to -0.30], Standard Error of Mean 0.0578

2. Secondary Outcome: Adjusted Mean Percentage Change From Baseline in Total Daily Insulin Dose at Week 24
Description: To compare the percent change from baseline in total daily insulin dose with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
Time Frame: Baseline and 24 weeks
Population: Number of subjects in full analysis set with non-missing baseline and at least one post-baseline value
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | DAPA 5 MG + INS | DAPA 10 MG + INS | PLA + INS
Number analyzed (Participants) | 270 | 267 | 266
Percentage change | -8.73 [-11.09 to -6.31] | -9.05 [-11.43 to -6.60] | 2.29 [-0.41 to 5.06]
Statistical Analysis 1: Comparison: DAPA 5 MG + INS vs PLA + INS; Difference vs. placebo in adjusted mean percentage change from baseline; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Adjusted for ln(baseline), treatment, week, randomization stratum, week*treatment, week*ln(baseline); Mean Difference (Final Values) = -10.78, 95% CI 2-sided [-13.73 to -7.72], Standard Error of Mean 1.5291
Statistical Analysis 2: Comparison: DAPA 10 MG + INS vs PLA + INS; Difference vs. placebo in adjusted mean percentage change from baseline; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Adjusted for ln(baseline), treatment, week, randomization stratum, week*treatment, and week*ln(baseline); Mean Difference (Final Values) = -11.08, 95% CI 2-sided [-14.04 to -8.02], Standard Error of Mean 1.5331

3. Secondary Outcome: Adjusted Mean Percentage Change From Baseline in Body Weight at Week 24
Description: To compare the percentage change from baseline in body weight with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
Time Frame: Baseline and 24 weeks
Population: Number of subjects in full analysis set with non-missing baseline and at least one post-baseline value
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | DAPA 5 MG + INS | DAPA 10 MG + INS | PLA + INS
Number analyzed (Participants) | 269 | 269 | 272
Percentage change | -3.22 [-3.76 to -2.69] | -3.76 [-4.29 to -3.22] | -0.02 [-0.57 to 0.54]
Statistical Analysis 1: Comparison: DAPA 5 MG + INS vs PLA + INS; Difference vs. placebo in adjusted mean percentage change from baseline; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Adjusted for ln(baseline), treatment, week, randomization stratum, week*treatment, and week*ln(baseline); Mean Difference (Final Values) = -3.21, 95% CI 2-sided [-3.96 to -2.45], Standard Error of Mean 0.3829
Statistical Analysis 2: Comparison: DAPA 10 MG + INS vs PLA + INS; Difference vs. placebo in adjusted mean percentage change from baseline; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Adjusted for ln(baseline), treatment, week, randomization stratum, week*treatment, and week*ln(baseline); Mean Difference (Final Values) = -3.74, 95% CI 2-sided [-4.49 to -2.99], Standard Error of Mean 0.3812

4. Secondary Outcome: Adjusted Mean Change From Baseline in 24-hour Continuous Glucose Monitoring (CGM) Mean Value at Week 24
Description: To compare the change from baseline in mean value of 24-hour glucose readings obtained from CGM with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
Time Frame: Baseline and 24 weeks
Population: The number of subjects in the full analysis set with non-missing baseline and at least one post-baseline value
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | DAPA 5 MG + INS | DAPA 10 MG + INS | PLA + INS
Number analyzed (Participants) | 252 | 255 | 257
mg/dL | -6.46 [-10.04 to -2.87] | -10.54 [-14.14 to -6.94] | 9.20 [5.57 to 12.83]
Statistical Analysis 1: Comparison: DAPA 5 MG + INS vs PLA + INS; Difference vs. placebo in adjusted mean change from baseline; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Adjusted for baseline, treatment, week, randomization stratum, week*treatment, and week*baseline; Mean Difference (Final Values) = -15.66, 95% CI 2-sided [-20.26 to -11.05], Standard Error of Mean 2.3468
Statistical Analysis 2: Comparison: DAPA 10 MG + INS vs PLA + INS; Difference vs. placebo in adjusted mean change from baseline; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Adjusted for baseline, treatment, week, randomization stratum, week*treatment, and week*baseline; Mean Difference (Final Values) = -19.74, 95% CI 2-sided [-24.34 to -15.14], Standard Error of Mean 2.3419

5. Secondary Outcome: Adjusted Mean Change From Baseline in 24-hour CGM Mean Amplitude of Glycemic Excursion (MAGE) Value at Week 24
Description: To compare the change from baseline in mean amplitude of glucose excursions (MAGE) of 24-hour glucose readings obtained from CGM with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
Time Frame: Baseline and 24 weeks
Population: Number of subjects in the full analysis set with non-missing baseline and at least one post-baseline value
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | DAPA 5 MG + INS | DAPA 10 MG + INS | PLA + INS
Number analyzed (Participants) | 252 | 255 | 257
mg/dL | -10.17 [-13.90 to -6.45] | -9.68 [-13.44 to -5.93] | -0.33 [-4.12 to 3.46]
Statistical Analysis 1: Comparison: DAPA 5 MG + INS vs PLA + INS; Difference vs. placebo in adjusted mean change from baseline; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Adjusted for baseline, treatment, week, randomization stratum, week*treatment, and week*baseline; Mean Difference (Final Values) = -9.85, 95% CI 2-sided [-14.66 to -5.03], Standard Error of Mean 2.4519
Statistical Analysis 2: Comparison: DAPA 10 MG + INS vs PLA + INS; Difference vs. placebo in adjusted mean change from baseline; Test type: Superiority; p = 0.0001, Mixed Models Analysis; Adjusted for baseline, treatment, week, randomization stratum, week*treatment, and week*baseline; Mean Difference (Final Values) = -9.36, 95% CI 2-sided [-14.16 to -4.55], Standard Error of Mean 2.4487

6. Secondary Outcome: Change From Baseline in the Percent of 24-hour Glucose Readings Obtained From CGM That Falls Within the Target Range of > 70 mg/dL and <= 180 mg/dL (%) at Week 24
Description: To compare the change from baseline in the percent of 24-hour glucose readings obtained from CGM that falls within the target range of >70 mg/dL and <=180 mg/dL with dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin after 24 weeks of double-blinded treatment
Time Frame: Baseline and 24 weeks
Population: Number of subjects in the full analysis set with non-missing baseline and at least one post-baseline value
Measure: Least Squares Mean (95% Confidence Interval); unit: % of readings
Arm/Group | DAPA 5 MG + INS | DAPA 10 MG + INS | PLA + INS
Number analyzed (Participants) | 252 | 255 | 257
% of readings | 5.92 [4.32 to 7.52] | 7.60 [5.98 to 9.21] | -3.10 [-4.73 to -1.47]
Statistical Analysis 1: Comparison: DAPA 5 MG + INS vs PLA + INS; Difference vs. placebo in adjusted mean change from baseline; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Adjusted for baseline, treatment, week, randomization stratum, week*treatment, and week*baseline; Mean Difference (Final Values) = 9.02, 95% CI 2-sided [6.97 to 11.06], Standard Error of Mean 1.0415
Statistical Analysis 2: Comparison: DAPA 10 MG + INS vs PLA + INS; Difference vs. placebo in adjusted mean change from baseline; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Adjusted for baseline, treatment, week, randomization stratum, week*treatment, and week*baseline; Mean Difference (Final Values) = 10.70, 95% CI 2-sided [8.66 to 12.74], Standard Error of Mean 1.0396

7. Secondary Outcome: Percentage of Subjects With HbA1c Reduction From Baseline to Week 24 Last Observation Carried Forward (LOCF) >= 0.5% and Without Severe Hypoglycemia Events at Week 24
Description: To compare dapagliflozin 5 mg or 10 mg plus adjustable insulin versus placebo plus adjustable insulin for the proportion of subjects achieving an HbA1c reduction from baseline to Week 24 visit >=0.5% without severe hypoglycemia events
Time Frame: Baseline and 24 weeks
Population: Number of subjects in the full analysis set with non-missing baseline and Week 24 (LOCF) values.
Measure: Count of Participants; unit: Participants
Arm/Group | DAPA 5 MG + INS | DAPA 10 MG + INS | PLA + INS
Number analyzed (Participants) | 266 | 267 | 269
Participants
  Number of Responders | 105 | 111 | 54
Statistical Analysis 1: Comparison: DAPA 5 MG + INS vs PLA + INS; Odds Ratio vs. Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic; Adjusted for baseline HbA1c and randomization strata; Odds Ratio (OR) = 2.71, 95% CI 2-sided [1.81 to 4.06], Standard Error of Mean 0.2058
Statistical Analysis 2: Comparison: DAPA 10 MG + INS vs PLA + INS; Odds Ratio vs. Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic; Adjusted for baseline HbA1c and randomization strata; Odds Ratio (OR) = 3.07, 95% CI 2-sided [2.05 to 4.60], Standard Error of Mean 0.2054

ADVERSE EVENTS:
Time Frame: All adverse events (AEs), including serious adverse events (SAEs), were collected from the time informed consent was signed throughout the treatment period (through week 24).
Arm/Group | DAPA 5 MG + INS | DAPA 10 MG + INS | PLA + INS
All-Cause Mortality (participants affected / at risk) | 0/271 | 0/270 | 0/272
Serious Adverse Events (participants affected / at risk) | 18/271 | 7/270 | 5/272
Other Adverse Events (participants affected / at risk) | 79/271 | 77/270 | 63/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAPA 5 MG + INS (N=271) | DAPA 10 MG + INS (N=270) | PLA + INS (N=272)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 7 (7) | 3 (3) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic hyperglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAPA 5 MG + INS (N=271) | DAPA 10 MG + INS (N=270) | PLA + INS (N=272)
Viral upper respiratory tract infection (Infections and infestations) | 39 (46) | 44 (56) | 42 (51)
Headache (Nervous system disorders) | 10 (11) | 15 (15) | 10 (11)
Pollakiuria (Renal and urinary disorders) | 22 (23) | 14 (15) | 6 (6)
Thirst (General disorders) | 6 (7) | 14 (14) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 16 (21) | 12 (12) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator requests permission to publish data from this study any such publication is to be agreed with AstraZeneca (AZ) in advance. The investigator agrees to provide AZ as soon as possible with drafts of proposed publications. Unless otherwise agreed, AZ shall have a period of 60 days from receipt of the proposed final manuscript to review it and may within such time require that submission for publication of the manuscript be delayed in order for AZ to file patent applications.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT02460978/SAP_000.pdf
  • Study Protocol (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT02460978/Prot_001.pdf